CLINICAL TRIAL: NCT02746861
Title: Web-based Training of Peers to Deliver Diabetes Self-Management Support
Brief Title: Peer-Supported Diabetes Self-Management Support
Acronym: DSMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: InquisitHealth, Inc. (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Ashwin Patel, Chief Medical Officer, InquisitHealth, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DSMS24; 5R43MD009555 (NIH)
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes
Keywords: peer mentor; peer supporter; peer coach; peer-to-peer mentoring
MeSH Terms: conditions — Diabetes Mellitus

ARMS (2):
- Diabetes Self-Management Support (DSMS) (Experimental): Patient receives 6-months of DSMS while receiving support from a trained peer mentor (Peer-supported DSMS).
  Interventions: Behavioral: Peer-Supported DSMS
- Usual Care (No Intervention): Patient continues to receive usual care.

INTERVENTIONS:
Behavioral: Peer-Supported DSMS — Phone, SMS/text, and smartphone-based intervention.
  Arms: Diabetes Self-Management Support (DSMS)

SUMMARY:
The objective is to evaluate the efficacy of a web-trained workforce of Hispanic and African American diabetes peer mentors delivering Diabetes Self-Management Support (DSMS) to patients with poorly-controlled diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* HbA1c>9%
* African American or Hispanic ethnicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Average reduction in HbA1c from baseline | 6-months

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin Patel, MD PhD, Principal Investigator — Chief Medical Officer
Locations (1):
- InquisitHealth, River Edge, New Jersey, United States